CLINICAL TRIAL: NCT00598910
Title: A Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Study to Investigate the Effect of Omacor (n-3 PUFA) on Lipid Parameters in HIV Infected Subjects Treated With HAART
Brief Title: Effect of Omacor on Triglycerides in HIV Infected Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was discontinued prematurely on December 18 2008 due to slow recruitment
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Joachim Luszick, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S185.4.001; 2007-001921-86
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Hyper-Triglyceridemia
Keywords: HIV infection
MeSH Terms: conditions — HIV Infections | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Omacor
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omacor — n-3 PUFA
  Arms: A
Drug: Placebo — Placebo
  Arms: B

SUMMARY:
Omacor is likely to decrease lipid parameters in HIV infected subjects. In these subjects the lipid are decrease due to HAART treatment

ELIGIBILITY:
Inclusion Criteria:

* Triglycerides between 200 and 800
* diagnosed HIV infection
* following HAART therapy

Exclusion Criteria:

* other malignant disease
* not compliant
* allergy against fish oil
* soy or olive oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percent change in serum triglycerides from baseline to treatment endpoint versus placebo | 12 weeks treatment

SECONDARY OUTCOMES:
Absolute change in serum triglycerides | 12 weeks
Absolute and percent change in cholesterol and cholesterol subfractions | 12 weeks
Absolute and percent change in apolipoprotein A and B | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (5):
- Germany (2):
  - Site 2, Bochum
  - Site 1, Hanover
- United Kingdom (3):
  - Site 3, London
  - Site 4, London
  - Site 5, London

REFERENCES:
- [Derived] Peters BS, Wierzbicki AS, Moyle G, Nair D, Brockmeyer N. The effect of a 12-week course of omega-3 polyunsaturated fatty acids on lipid parameters in hypertriglyceridemic adult HIV-infected patients undergoing HAART: a randomized, placebo-controlled pilot trial. Clin Ther. 2012 Jan;34(1):67-76. doi: 10.1016/j.clinthera.2011.12.001. Epub 2011 Dec 31. PMID 22212377